CLINICAL TRIAL: NCT02176343
Title: Retrospective / Prospective Clinical Study of AcrySof® IQ ReSTOR® +2.5 D Multifocal Toric Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-14-005
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-05

CONDITIONS: Cataract; Presbyopia; Corneal Astigmatism
Keywords: Cataract; Intraocular lens; ACRYSOF IQ ReSTOR + 2.5 D Multifocal Toric IOL
MeSH Terms: conditions — Cataract; Presbyopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ReSTOR Toric +2.5 (Experimental): AcrySof® IQ ReSTOR® +2.5 D Multifocal Toric IOL previously implanted during cataract surgery
  Interventions: Device: AcrySof® IQ ReSTOR® +2.5 D Multifocal Toric IOL

INTERVENTIONS:
Device: AcrySof® IQ ReSTOR® +2.5 D Multifocal Toric IOL — Multifocal IOL with extended secondary focal point and astigmatism correction implanted for long-term use over the lifetime of the cataract patient
  Other Names: Model SV25T2; Model SV25T3; Model SV25T4; Model SV25T5

SUMMARY:
The purpose of this study is to characterize the safety and effectiveness of the ACRYSOF IQ ReSTOR +2.5 diopter (D) Multifocal Toric Intraocular Lens (IOL) in subjects at least 3 months and no more than 14 months after IOL implantation.

DETAILED DESCRIPTION:
This is a retrospective and prospective clinical study comprised of a retrospective chart review for preoperative, surgical and early postoperative data, and a prospective postoperative visit conducted at least 3 months but not more than 14 months after IOL implantation.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form and be willing to come in for a visit at least 3 months and not more than 14 months after IOL implantation with the AcrySof® IQ ReSTOR® +2.5 D Multifocal Toric IOL (Models SV25T2, SV25T3, SV25T4 and SV25T5);
* Must be implanted with the correct lens based on preoperative corneal astigmatism as specified in the protocol;
* Must complete a visit within 10 days after IOL implantation;
* Successful capsular bag implantation with no surgical complications;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* IOL implanted prior to the AcrySof® IQ ReSTOR® +2.5 D Multifocal Toric IOL;
* Ocular or intraocular infection or inflammation at the time of the preoperative visit;
* Any ocular surgery or intraocular laser procedure at or prior to the surgical visit;
* Any conditions affecting the cornea (eg. corneal dystrophy, severe dry eye) at the preoperative visit;
* Retinal conditions (e.g. degenerative retinal conditions, history of retinal detachment, diabetic retinopathy) at the preoperative visit;
* Known history of Type 1 or 2 diabetes for more than 5 years;
* Any ocular or systemic co-morbidity at the preoperative visit;
* Pregnant at the preoperative visit or at the time of Postoperative Visit 2;
* Preoperative corneal astigmatism ≤ 0.50 D;
* Participation in another clinical study at the preoperative visit or at the time of the final study visit;
* Other protocol-specified exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2014-08-22 (Actual); Study Completion 2014-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, GCRA, Surgical, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 study centers located in Australia.
Pre-assignment Details: Of the 37 enrolled, 6 subjects were exited as screen failures and were ineligible to participate in the study. This reporting group includes all subjects who provided informed consent and were determined to be eligible based upon the inclusion and exclusion criteria (As Treated) (31).
Groups:
- ReSTOR Toric +2.5: AcrySof® IQ ReSTOR® +2.5 D Multifocal Toric Intraocular Lens (IOL)
Period: Overall Study
Arm/Group | ReSTOR Toric +2.5
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: As Treated
Groups:
- ReSTOR Toric +2.5: AcrySof® IQ ReSTOR® +2.5 D Multifocal Toric IOL
Arm/Group | ReSTOR Toric +2.5
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Reduction in Cylinder
Description: Manifest refraction cylinder was measured monocularly (each eye separately) with best correction (phoropter or trial lenses) under photopic (well-lit) lighting conditions using a 100% contrast ETDRS chart at 4 meters (m) from the subject. Percent reduction in cylinder was calculated as the difference between the postoperative magnitude of manifest refractive cylinder and the preoperative magnitude of keratometric cylinder divided by the intended reduction in cylinder [defined as the difference between the intended (from toric calculator) magnitude of the postoperative manifest refractive cylinder and the preoperative keratometric cylinder], multiplied by 100%. One eye (primary eye) contributed to the analysis.
Time Frame: Preoperative and Postoperative Visit (3 to 14 months after IOL implantation)
Population: As Treated
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ReSTOR Toric +2.5
Number analyzed (Participants) | 31
percent change | 60.94 (38.17)

2. Primary Outcome: Percentage of Subjects With Manifest Refraction Cylinder ≤ 0.50 D
Description: Manifest refraction cylinder was measured monocularly with best correction under photopic lighting conditions using a 100% contrast ETDRS chart at 4 m from the subject. One eye (primary eye) contributed to the analysis.
Time Frame: Preoperative and Postoperative Visit (3 to 14 months after IOL implantation)
Population: As Treated
Measure: Number; unit: percentage of subjects
Arm/Group | ReSTOR Toric +2.5
Number analyzed (Participants) | 31
percentage of subjects | 67.7

3. Primary Outcome: Percentage of Subjects (With Preoperative Astigmatism > 1.00 D) With Manifest Refraction Cylinder ≤ 1.00 D
Description: as for outcome 2
Time Frame: Preoperative and Postoperative Visit (3 to 14 months after IOL implantation)
Population: This analysis population includes all subjects who provided informed consent and were determined eligible based upon the inclusion and exclusion criteria, having preoperative astigmatism > 1.00 D.
Measure: Number; unit: percentage of subjects
Arm/Group | ReSTOR Toric +2.5
Number analyzed (Participants) | 12
percentage of subjects | 100.0

4. Primary Outcome: Mean Uncorrected Distance Visual Acuity
Description: Visual Acuity (VA) was tested monocularly without visual correction under photopic (well-lit) conditions using a 100% contrast ETDRS chart positioned 4 m from the subject. A +0.25 D spherical power additional lens was used to correct for optical infinity. VA was measured in logMAR (logarithm of the minimum angle of resolution), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity. One eye (primary eye) contributed to the analysis.
Time Frame: Preoperative and Postoperative Visit (3 to 14 months after IOL implantation)
Population: As Treated
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric +2.5
Number analyzed (Participants) | 31
logMAR | 0.07 (0.12)

5. Primary Outcome: Mean Uncorrected Near Visual Acuity
Description: VA was tested monocularly without visual correction under photopic lighting conditions using a 100% contrast near ETDRS chart set at 40 cm on the nearpoint rod of the phoropter. VA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity. One eye (primary eye) contributed to the analysis.
Time Frame: Preoperative and Postoperative Visit (3 to 14 months after IOL implantation)
Population: As Treated
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric +2.5
Number analyzed (Participants) | 31
logMAR | 0.38 (0.16)

6. Primary Outcome: Mean Uncorrected Intermediate Visual Acuity
Description: VA was tested monocularly without visual correction under photopic lighting conditions using a 100% contrast near ETDRS chart set at 53 cm on the nearpoint rod of the phoropter. VA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity. One eye (primary eye) contributed to the analysis.
Time Frame: Preoperative and Postoperative Visit (3 to 14 months after IOL implantation)
Population: As Treated
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric +2.5
Number analyzed (Participants) | 31
logMAR | 0.25 (0.16)

7. Primary Outcome: Mean Best Corrected Distance Visual Acuity (BCDVA)
Description: VA was tested monocularly with best correction under photopic lighting conditions using a 100% contrast ETDRS chart at 4 m away from the subject. VA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity. One eye (primary eye) contributed to the analysis.
Time Frame: Preoperative and Postoperative Visit (3 to 14 months after IOL implantation)
Population: As Treated
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric +2.5
Number analyzed (Participants) | 31
logMAR | -0.03 (0.08)

8. Primary Outcome: Mean IOL Rotation
Description: Lens axis orientation (position of the lens within the capsular bag) as indicated by indentations on the IOL was assessed during slit lamp examination. IOL rotation (the difference between the achieved lens axis orientation at visit and achieved axis placement at surgery) was measured in degrees. One eye (primary eye) contributed to the analysis.
Time Frame: Preoperative and Postoperative Visit (3 to 14 months after IOL implantation)
Population: As Treated
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | ReSTOR Toric +2.5
Number analyzed (Participants) | 31
degrees | 3.74 (3.86)

ADVERSE EVENTS:
Time Frame: The time period of collection of AEs was preoperative to postoperative visit 3-14 months after IOL implantation. This analysis population includes all subjects who provided informed consent and were determined eligible based upon inclusion and exclusion criteria (As Treated).
Description: An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational product. AEs were obtained as solicited and volunteered comments from subjects and as observations by the study Investigator as outlined in the study protocol.
Groups:
- ReSTOR Toric +2.5: All subjects implanted with AcrySof® IQ ReSTOR® +2.5 D Multifocal Toric IOL
Arm/Group | ReSTOR Toric +2.5
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 4/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReSTOR Toric +2.5 (N=31)
Macular oedema (Eye disorders) | 1
Retinal vein occlusion (Eye disorders) | 1
Strabismus (Eye disorders) | 1
Staphylococcal infection (Infections and infestations) | 1
Intra-ocular injection (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ReSTOR Toric +2.5 (N=31)
Photopsia (Eye disorders) | 2
Knee arthroplasty (Surgical and medical procedures) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.